CLINICAL TRIAL: NCT03608371
Title: Phase 2A, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BTRX-246040 in Parkinson's Disease Subjects With Motor Fluctuations
Brief Title: BTRX-246040 Study in Participants With Parkinson's Disease With Motor Fluctuations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BlackThorn Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEP-PD-201
Record Dates: First submitted 2018-05-09; First posted 2018-07-31 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease; Motor Disorder
MeSH Terms: conditions — Parkinson Disease; Motor Disorders

STUDY DESIGN:
Intervention Model Description: The study consists of 3 sequential, single ascending dose cohorts of 8 participants each with a 6:2 randomization to BTRX-246040 or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BTRX-246040 Cohort 1 (Experimental): BTRX-246040 40 mg administered orally
  Interventions: Drug: BTRX-246040
- BTRX-246040 Cohort 2 (Experimental): BTRX-246040 80 mg administered orally
  Interventions: Drug: BTRX-246040
- BTRX-246040 Cohort 3 (Experimental): BTRX-246040 120 mg administered orally
  Interventions: Drug: BTRX-246040
- Placebo Cohorts 1-3 (Placebo Comparator): Placebo is administered orally at the same number of capsules as active drug in each Cohort. Placebo capsules consist of inactive ingredients and look identical to BTRX-246040.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BTRX-246040 — oral capsule
  Arms: BTRX-246040 Cohort 1; BTRX-246040 Cohort 2; BTRX-246040 Cohort 3
Drug: Placebo — oral capsule matching BTRX-246040 capsule
  Arms: Placebo Cohorts 1-3

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and efficacy of BTRX-246040 in participants with Parkinson's Disease who have motor fluctuations and predictable early morning off periods.

DETAILED DESCRIPTION:
Study treatment is 1 day and total duration of the study is up to 36 days, including an approximate 28-day screening period. The study consists of 3 sequential, ascending dose cohorts of 8 participants each with a 6:2 randomization to BTRX-246040 or placebo. The planned dosing for each cohort is 40, 80, and 120 mg. After enrollment of the first cohort is completed, doses for subsequent cohorts may be modified based on review of the available data (safety, tolerability, efficacy, and pharmacokinetics) by an unblinded Dosing Review Committee (DRC). A similar review and determination of dosing for the subsequent cohort is to be performed after completion of each cohort and based on all data available from previous cohorts.

Participants who meet entry criteria assessed at the screening visit (up to 28 days prior to Day 1) present to the clinic on the morning of Day 1 (treatment day) in the practically defined OFF state (having withheld anti-parkinsonian medications after 10:00 PM the evening prior). Participants are to be dosed with study drug and remain on site for an 8-hour observation period with Unified Parkinson's Disease Rating Scale (UPDRS) Part III motor response, dyskinesia rating and ON/OFF status assessed pre-dose, every 30 minutes for 4 hours post-dose, and then hourly for 4 additional post-dose hours (i.e., 8 hours total post-dose) prior to being discharged. Blood for pharmacokinetics are to be collected 6 times at scheduled intervals within the 8-hour observation period. A follow-up safety visit is scheduled 7 days later.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease (PD), consistent with the United Kingdom PD Society Brain Bank Criteria for the Diagnosis of PD
* Men or women ≥ 30 years old and ≤ 76 years old
* Female participants must be either surgically sterilized or 2 years post menopausal at screening
* Modified Hoehn and Yahr Staging ≤ 3 in the ON state
* Montreal Cognitive Assessment (MoCA) Score ≥ 26
* Currently has a clear and decisive response to levodopa, and receiving a stable dose of levodopa (at least 4 doses per day of levodopa or ≥ 3 doses per day of RytaryTM (carbidopa and levodopa) extended-release capsules for at least 4 weeks prior to screening)
* Experiencing motor fluctuations during waking hours with at least 2 hours of OFF periods each day, including predictable early morning OFF periods, based on participant assessment
* Able to participate in the study in the practically defined OFF state
* All anti-parkinsonian medications maintained at a stable dose for at least 4 weeks prior to the initial Screening Visit with the exception of monoamine oxidase B (MAO-B) inhibitors, which must be maintained at a stable level for at least 8 weeks prior to the screening visit
* Approved by a central Enrollment Authorization Committee as meeting entry criteria and being a suitable candidate for the study
* Male participants agree to use a reliable method of birth control during the study and for at least 90 days following the last dose of BTRX-246040 or placebo
* Informed and given ample time and opportunity to think about his/her participation in this study and has given his/her written informed consent on an Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved consent form
* Judged to be reliable and able to keep all appointments for clinic visits, tests, and procedures, including venipuncture, and examinations required by the protocol

Exclusion Criteria:

* Diagnosis of secondary or an atypical Parkinsonian syndrome
* Severe disabling dyskinesia
* Clinically significant psychosis or hallucinations or history of psychosis in past 6 months
* History of previous neurosurgery for PD
* Currently or previously on Duopa/Duodopa
* Currently taking apomorphine
* Has a diagnosis or history of a substance related disorder per Diagnostic and Statistical Manual of Mental Disorders V edition (DSM-V) criteria (including alcohol but excluding nicotine and caffeine), during the 12 months prior to the Screening Visit
* Medical or recreational use of marijuana in the 6 months prior to the Screening Visit
* Has tested positive at the Screening Visit for drugs of abuse (opiates, cannabinoids, methadone, cocaine, and amphetamines [including ecstasy])
* Active suicidal ideation within 1 year prior to the Screening Visit as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the Columbia- Suicide Severity Rating Scale (C-SSRS) or attempted suicide within the last 1 year
* Current major depressive episode or a Beck Depression Inventory-II (BDI-II) score above 19. Participants receiving treatment for depression with antidepressants may be enrolled if they have been on a stable daily dose for at least 8 weeks before the Screening Visit and are clinically stable in the opinion of the Principal Investigator
* Currently or within 8 weeks of screening receiving bupropion
* Exposure to neuroleptics (antipsychotic drugs) for more than 1 month within the past 2 years, or any exposure within the past year
* Any malignancy in the 5 years prior to randomization (excluding successfully treated basal cell carcinoma of the skin or cervical carcinoma in situ)
* Current or previous diagnosis of malignant melanoma or the presence of any suspicious skin lesion based on physical exam findings
* Any other clinically significant medical condition or circumstance prior to randomization that, in the opinion of the Investigator, could affect participant safety, preclude evaluation of response, interfere with the ability to comply with study procedures, or prohibit completion of the study (e.g., uncontrolled diabetes mellitus, renal or hepatic impairment, coronary artery disease, evidence of significant active cardiac, respiratory, or hematologic disease, cancer with < 5 year remission (excluding successfully treated basal cell carcinoma of the skin or cervical carcinoma in situ), chronic pain, fibromyalgia or gastric bypass)
* Prior seizures (other than childhood febrile seizure) or other condition that would place the participant at increased risk of seizures or is taking anticonvulsants for seizure control
* History of serious head injury (e.g., skull fracture, cerebral contusion, or trauma resulting in prolonged unconsciousness), intracranial neoplasm or hemorrhage
* Orthostatic hypotension that is symptomatic or requires medication
* Participation in another study of an investigational medicinal product (IMP) or medical device currently or in the last 30 days or within 5 half-lives of the IMP (whichever is longer) prior to Screening
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels ≥ 2x upper limit of normal (ULN) or glomerular filtration rate ≤ 60 mL/min at Visit 1 (screening)
* Nephritic syndrome, end-stage renal disease (and using renal replacement therapy such as hemodialysis or peritoneal dialysis), or a serum creatinine ≥ 2 mg/dL (≥ 172 μmol/L) at the Screening Visit
* Any other clinically significant abnormalities (i.e., laboratory deviations requiring acute medical intervention or further medical evaluation) in laboratory results at screening including clinical chemistries, hematology, and urinalysis, that, in the judgment of the Investigator, should preclude a participant's participation at study entry
* Electrocardiogram (ECG) abnormalities at Visit 1 (screening) or Visit 2 that, in the judgment of the Investigator, are clinically significant related to the participant's participation
* Using the following concomitant medications (contact the Sponsor-designated medical monitor to determine eligibility when in doubt):

  1. proton pump inhibitors within 5 half-lives of Screening
  2. fluoxetine and irreversible monoamine oxidase inhibitors within 4 weeks of Screening
* Currently taking or have taken, within 5 half-lives of Screening, any medications or supplements that are strong inhibitors or inducers of CYP3A4
* A known hypersensitivity to gelatin capsules
* Investigator site personnel directly affiliated with this study, and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Employees of the Sponsor or of any third-party organizations involved in study who require exclusion of their employees
* Have participated in a clinical trial or any other type of medical research judged by the Investigator to be scientifically or medically incompatible with this study within 30 days prior to Visit 1 (screening)
* Previous completion or withdrawal from this study or any other study investigating BTRX-246040 (previously called LY2940094)

Ages: 30 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane M Tiller, M.D., Study Director — BlackThorn Therapeutics, Inc. (Sponsor)
Locations (4):
- United States (4):
  - BlackThorn Investigator Site, Hallandale, Florida
  - BlackThorn Investigator Site, Farmington Hills, Michigan
  - BlackThorn Investigator Site, Durham, North Carolina
  - BlackThorn Investigator Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo administered orally at the same number of capsules as active drug in each Cohort
Period: Overall Study
Arm/Group | BTRX-246040 Cohort 1 | BTRX-246040 Cohort 2 | BTRX-246040 Cohort 3 | Placebo
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BTRX-246040 Cohort 1 | BTRX-246040 Cohort 2 | BTRX-246040 Cohort 3 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 62.3 (7.09) | 60.5 (8.07) | 63.5 (4.76) | 66.3 (5.35) | 63.15 (6.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 2 | 14
  Male | 3 | 1 | 2 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 0 | 1 | 6
  Not Hispanic or Latino | 1 | 6 | 6 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 6 | 6 | 5 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Maximal Change in UPDRS Part III From Predose to Postdose on Day 1
Description: UPDRS = Unified Parkinson's Disease Rating Scale. The Unified Parkinson's Disease Rating Scale (UPDRS) Part III is a 14-item rating scale, which consists of the motor examination. Each item is scored from 0 (Normal) to 4 (Most severe). The score ranges from 0-56.
Time Frame: From pre-dose to 8 hours post-dose on Day 1
Population: Modified Intent to Treat (mITT): all randomized participants who received at least 1 dose of the investigational product and had at least 1 post-baseline scoring of motor activity.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Combined BTRX-246040: Combined BTRX-246040 groups
Arm/Group | BTRX-246040 Cohort 1 | BTRX-246040 Cohort 2 | BTRX-246040 Cohort 3 | Combined BTRX-246040 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 18 | 6
score on a scale | -22.0 (7.01) | -12.5 (4.68) | -11.2 (3.92) | -15.2 (7.08) | -17.0 (12.07)

2. Secondary Outcome: Duration of ON Time on Day 1
Description: ON is the typical functional state when patients are receiving medication and have a good response.
  OFF is the typical functional state when patients have a poor response in spite of taking medications.
Time Frame: From dose to 8 hours post-dose on Day 1
Population: Modified Intent to Treat (mITT): all randomized participants who received at least 1 dose of the investigational product and had at least 1 post-baseline scoring of motor activity. 21 participants reached an ON status on Day 1; however, only 12 participants had a time recorded for when they reached OFF status on Day 1. Therefore, Duration of ON Time on Day 1 is only available for 12 participants.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BTRX-246040 Cohort 1 | BTRX-246040 Cohort 2 | BTRX-246040 Cohort 3 | Combined BTRX-246040 | Placebo
Number analyzed (Participants) | 3 | 4 | 1 | 8 | 4
hours | 2.983 (1.8144) | 3.750 (1.8484) | 4.000 | 3.494 (1.6095) | 4.250 (1.5000)

3. Secondary Outcome: Percentage of Participants Who Turned ON on Day 1
Description: as for outcome 2
Time Frame: From dose to 8 hours post-dose on Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BTRX-246040 Cohort 1 | BTRX-246040 Cohort 2 | BTRX-246040 Cohort 3 | Combined BTRX-246040 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 18 | 6
Participants | 6 | 6 | 4 | 16 | 5

4. Secondary Outcome: Time to ON on Day 1
Description: as for outcome 2
Time Frame: From dose to 8 hours post-dose on Day 1
Population: Modified Intent to Treat (mITT): all randomized participants who received at least 1 dose of the investigational product and had at least 1 post-baseline scoring of motor activity. 21 participants reached an ON status on Day 1.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BTRX-246040 Cohort 1 | BTRX-246040 Cohort 2 | BTRX-246040 Cohort 3 | Combined BTRX-246040 | Placebo
Number analyzed (Participants) | 6 | 6 | 4 | 16 | 5
hours | 3.575 (2.7749) | 2.583 (2.7462) | 3.646 (2.7742) | 3.221 (2.6231) | 3.200 (2.8417)

5. Secondary Outcome: Area Under the Curve for UPDRS Part III During the 8 Hours of Assessment on Day 1
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) Part III is a 14-item rating scale, which consists of the motor examination. Each item is scored from 0 (Normal) to 4 (Most severe). UDPRS Part III was assessed pre-dose and every 30 minutes for 4 hours and then hourly for another 4 hours (i.e., 8 hours following study drug administration) on Day 1.
Time Frame: From pre-dose to 8 hours post-dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*minutes
Arm/Group | BTRX-246040 Cohort 1 | BTRX-246040 Cohort 2 | BTRX-246040 Cohort 3 | Combined BTRX-246040 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 18 | 6
score on a scale*minutes | 20224.50 (2301.418) | 15464.33 (5214.729) | 11682.42 (2231.434) | 15790.42 (4894.202) | 17547.08 (3110.784)

6. Secondary Outcome: Change From Pre-dose Dyskinesia Rating (From the UPDRS Part III Motor Response and Dyskinesia Assessment)
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) Part III is a 14-item rating scale, which consists of the motor examination. Each item is scored from 0 (Normal) to 4 (Most severe). An additional single item to rate dyskinesia was added to the UDPRS and was rated from 0 (no dyskinesia) to 4 (severe dyskinesia: maximal amplitude and present during most of the examinations).
Time Frame: From pre-dose to 8 hours post-dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BTRX-246040 Cohort 1 | BTRX-246040 Cohort 2 | BTRX-246040 Cohort 3 | Combined BTRX-246040 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 18 | 6
score on a scale
  Postdose Day 1 Change, 30 minutes postdose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Postdose Day 1 Change, 60 minutes postdose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Postdose Day 1 Change, 90 minutes postdose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Postdose Day 1 Change, 120 minutes postdose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Postdose Day 1 Change, 150 minutes postdose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Postdose Day 1 Change, 180 minutes postdose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Postdose Day 1 Change, 210 minutes postdose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Postdose Day 1 Change, 240 minutes postdose | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Postdose Day 1 Change, 5 hours postdose | 0.3 (0.82) | 0.0 (0.00) | 0.0 (0.00) | 0.1 (0.47) | 0.0 (0.00)
  Postdose Day 1 Change, 6 hours postdose | 0.3 (0.82) | 0.0 (0.00) | 0.3 (0.52) | 0.2 (0.55) | 0.0 (0.00)
  Postdose Day 1 Change, 7 hours postdose | 0.3 (0.82) | 0.0 (0.00) | 0.2 (0.41) | 0.2 (0.51) | 0.0 (0.00)
  Postdose Day 1 Change, 8 hours postdose | 0.0 (0.00) | 0.0 (0.00) | 0.2 (0.41) | 0.1 (0.24) | 0.0 (0.00)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 8 (+/- 1 day) or Early Termination visit, an average of 7 days.
Description: All participants received study drugs and were monitored for AEs through Day 8 (+/- 1 day) or Early Termination Visit. The Investigators were responsible for following adverse event through to resolution.
Arm/Group | BTRX-246040 Cohort 1 | BTRX-246040 Cohort 2 | BTRX-246040 Cohort 3 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 3/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BTRX-246040 Cohort 1 (N=6) | BTRX-246040 Cohort 2 (N=6) | BTRX-246040 Cohort 3 (N=6) | Placebo (N=6)
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0
Blood pressure systolic decreased (Investigations) | 0 | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 0 | 0
Urine ketone body present (Investigations) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT03608371/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT03608371/SAP_001.pdf